CLINICAL TRIAL: NCT06616129
Title: Preoperative RIsk Assessment and Shared Decision-Making in Patients Eligible for Cardiac Surgery (PRIME-study): a Study Protocol for a Single Center Non-randomized Prospective Trial
Brief Title: A Study Protocol for Research Investigating How Geriatric Risk Assessment and Shared Decision-making Conversations Affect Treatment Decisions and Quality of Life in Patients Eligible for Open-heart Surgery.
Acronym: PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Hanze University of Applied Sciences Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RR number: 202100724
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Frail Elderly Persons; Cardiac Surgery
Keywords: cardiothoracic surgery; decision-making; quality of life; frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRIME-Group (Experimental)
  Interventions: Diagnostic Test: Geriatric assessment; Other: Shared decision-making conversation
- Control Group (No Intervention)

INTERVENTIONS:
Diagnostic Test: Geriatric assessment — At the clinic further information on the somatic, social, psychological and functional domain will be gathered by the nurse and two validated tests to map the vulnerability and resilience of the patient will be used; the Cognitive Impairment Test and the timed Up and Go Test.
  Arms: PRIME-Group
Other: Shared decision-making conversation — The nurse and nurse practitioner together will talk with the patient and their partner about possible treatment options as well as patients' expectations, preferences and their life in general.
  During the conversation the OPT (Outcome Prioritization Tool) will be used to clarify the most important goals of treatment for the patient. The OPT exists of four universal treatment goals rated on a visual analogue scale from 0 to 100. The goals represented are: life extension, maintaining independence, reducing pain and reducing other symptoms. The goals will be explained and the patient will be asked to rate each outcome according to the trade-off principle meaning that two outcomes cannot be rated equally.
  Arms: PRIME-Group

SUMMARY:
The goal of this study is to determine whether intervention by the PRIME clinic influences cardiac treatment decisions, as well as patients quality of life and healthcare utilization.

The main questions this study aims to answer are:

* Does PRIME consultation influence treatment recommendations?
* Does a personalized treatment plan for cardiac patients influence health-related quality of life?
* Does a personalized treatment plan influence healthcare costs (in terms of quality-adjusted life years)?

Participants will:

* Visit the PRIME clinic once
* Complete quality of life questionnaires twice
* Track their healthcare usage over the course of a year and complete a corresponding questionnaire four times.

DETAILED DESCRIPTION:
The primary outcome of this study is the difference between treatment recommendations; the first treatment recommendation (the decision before the patient visits the outpatient clinic) will be compared with the treatment recommendation after the assessment at the outpatient clinic.

Secondary and other outcomes that will be collected are baseline demographic data including age, gender, body mass index, education level, European System for Cardiac Operative Risk Evaluation II (EuroSCORE II) and co-morbidities such as stroke, reduced cognitive function, chronic obstructive pulmonary disease (COPD) GOLD III or IV, renal failure (a reduced renal function prior to surgery with a kreatinine level ≥150mmol/L), a reduced left ventricular function, reduced mobility, cardiac reoperation and type of surgical procedure (CABG, valve replacement or repair, surgery of the thoracic aorta or a combination of several procedures).

Data will be collected using several questionnaires:

* Health-related Quality of Life (the RAND-36 questionnaire)
* The Katz Index of Independence in Activities of Daily Living to assess functional status
* The Cognitive Impairment Test
* The Timed Up and Go Test
* Outcome Prioritization Tool to assess the most important goals of treatment The RAND-36 and KATZ-ADL will be completed by all patients, including those receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and older
* Eligible for cardiac surgery
* Having two or more risk factors: stroke; reduced cognitive function; Chronic Obstructive Pulmonary Disease (COPD); obesity; reduced left ventricular ejection fraction; renal failure; reduced mobility; cardiac reoperation; and the complexity of the procedure.

Exclusion Criteria:

* Unable to read or understand Dutch

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference between the treatment recommendation provided by the multidisciplinary Heart Team prior to the patients visit to the PRIME-clinic and the treatment advice from the Heart Team after the patients visit to the PRIME-clinic. | From enrollment to the second treatment advice of the heart team, typically within 8 weeks. .
  After the patient is referred to the UMCG, the patients situation is discussed by the heart team, resulting in a treatment recommendation, which is documented in the electronic patient record. If the patient meets the inclusion criteria for the PRIME-study, they will also be invited to the PRIME-clinic (usually within a week). The findings from the PRIME-clinic are then discussed the same day during the heart team meeting, after which a treatment recommendation is formulated again.
  A difference in treatment recommendation is noted when the initial recommendation is revised, opting for a less invasive or conservative treatment instead of open-heart surgery.

SECONDARY OUTCOMES:
Health related quality of life, SF-36 | From enrollment to one year after
  Health-related quality of life is measured using the validated SF-36 questionnaire, which consists of 36 items that assess eight health dimensions: physical functioning, role limitations due to physical health issues, role limitations due to emotional problems, social functioning, emotional well-being, energy levels and fatigue, pain, and overall perceptions of general health. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health. Two composite scores can be derived from these domains: the Physical Component Score and the Mental Component Score.
The cost-effectiveness ratio, an analysis that combines both the EQ-5D-5L (for health gains) and the Medical Cost Questionnaire (for costs) | From enrollment to one year after
  Both the MCQ and EQ-5D-5L will be administered at 3, 6, 9, and 12 months following the PRIME-clinic visit.
  The MCQ will be used to measure the healthcare utilization. This includes both direct medical costs (such as hospitalizations, medication, and treatments) as well as indirect costs (such as productivity losses). Additionally, Quality-Adjusted Life Years (QALYs) are calculated using the EQ-5D-5L, which measures health-related quality of life.
  Using these data (QALYs and costs), the cost per QALY is calculated, representing the ratio between the costs of treatment and the health gains achieved. A lower cost per QALY indicates that the treatment is more cost-effective.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. Mariani, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will make the dataset available once all data has been anonymized.
Supporting Information: Study Protocol
Time Frame: The protocol will be made available after it has been published.
Access Criteria: The data will be available on reasonable request.